

#### INFORMED VOLUNTARY CONSENT FORM

Document Code: ÜNV-GOAEK-FRM-002

Release Date: 17.09.2019

Revision No: 03

Revision Date: 01.06.2022


**STUDY TITLE:** The effect of the use of digital games on learning satisfaction and self-confidence in providing nursing students with the ability to apply subcutaneous injections.

You are asked to participate in a research study, the information of which is listed below. The decision whether or not to participate in the study is entirely yours. Before deciding whether or not you want to participate, it's important to understand why the research is being done, how your information will be used, what the study involves, the possible benefits and risks, or aspects that may cause inconvenience. Please take the time to read the following information carefully. If you decide to participate in the study, **sign the Study Participation**Consent Form. You are free to leave the study at any time. No payment will be made to you for participating in the Work or you will not be asked to contribute any material/material contributions. All materials to be used in the research and all expenses that can be made will be covered by the researcher.

#### SUBJECT AND PURPOSE OF THE STUDY

Skills laboratory training in nursing education is very important in teaching basic skills of nursing. One of the basic nursing skills taught in laboratory practice is drug practice. Medication is one of the practitioner roles of the nurse and ensuring patient safety is the most important principle in this practice. Therefore, on the nurse's medication management; must be competent in the preparation of drugs, their correct and safe administration, patient education and monitoring of the desired effects and side effects of drugs. Subcutaneous drug administration, which is one of the parenteral drug administration methods, and drugs such as heparin, horman, vaccine and insulin are applied. In order to increase the psychomotor skills of nursing students, innovative approaches and educational technologies such as reality augmented simulation models, virtual reality applications and haptic systems and computer-aided education (BDE) are needed. Computer-aided education; It is defined as the provision of education through information and communication technologies. One of the computer-aided education methods frequently used today is educational digital game software. These types of software enable the student to actively participate in the learning process and develop psychomotor skills. Digital games have been reported to improve cognitive skills in learning, increase information processing speed, improve reaction time, and improve attention skills such as visual-spatial attention. Based on the hypothesis that it improves health knowledge, skills and behavior, reduces the anxiety level of the student and increases learning satisfaction, in this research, the effect of a digital game-based application on learning satisfaction and self-confidence will be determined in the acquisition of the ability of subcutaneous drug application by nursing students.

## **WORKING OPERATIONS**

No attempt will be made to harm you during the working time. If you agree to participate in the study, you will be randomly assigned to the experimental or control group. In the meantime, you will fill out the "Student Information Form" developed by the researchers and consist of 8 questions and you will use the "Subcutaneous Injection



#### INFORMED VOLUNTARY CONSENT FORM

Document Code: ÜNV-GOAEK-FRM-002

Release Date: 17.09.2019

Revision No: 03

Revision Date: 01.06.2022


Information Test". If you take part in the experimental group, after the theoretical part of the subcutaneous injection application in the curriculum is completed, you will play the digital game prepared for the subcutaneous injection application offered to you for a week and then you will apply the subcutaneous injection process on low realistic arm / abdomen models in the subcutaneous injection application laboratory course in the curriculum. During the subcutaneous injection application, you will be evaluated by the researcher with the "Subcutaneous Injection Application Skill Checklist". After the application, you will fill out the "Student Satisfaction and Self-Confidence in Learning Scale" consisting of 13 items and answer the "Subcutaneous Injection Knowledge Test" again. If you take part in the control group, all the steps counted in the experimental group will be applied to you, but you will not play the digital game prepared for the application. It will take you an estimated 5-10 minutes to complete the questionnaires and scales.

### WHAT ARE THE BENEFITS OF TAKING PART IN THE STUDY?

The education you receive as students of the Department of Nursing consists of theoretical, laboratory and clinical practice sections and your basic nursing skills begin to develop from the first year. However, the application of invasive interventions by nursing students in terms of patient safety in the clinical field may pose a number of risks. Today, especially the use of digital-based educational games offered by technology allows students to develop basic nursing skills without risking patient safety. For this reason, by participating in this study, you will help determine the effect of a digital game-based application on learning satisfaction and self-confidence in the acquisition of subcutaneous drug administration skills and contribute to the literature.

### WHAT IS THE COST OF PARTICIPATING IN THIS STUDY?

You will not be burdened financially by participating in the Study and you will not be paid.

## SHOULD I PARTICIPATE IN THE STUDY?

Whether or not to take part in this work is entirely up to you. Even if you sign this form right now, you are free to stop working at any time without giving a reason.

#### HOW WILL MY PERSONAL INFORMATION BE USED?

Your study researcher will use your personal information to conduct the research and statistical analysis, but your personally identifiable information will be kept confidential. Only if necessary, ethics committees or official authorities can review information about you. At the end of the study, you have the right to ask for information about your own results. The results of the study may be published in the medical literature at the end of the study, but your identity will not be disclosed.

## **CONTACT PERSONS FOR QUESTIONS AND PROBLEMS:**

NAME : Burcu DEMİRCAN

JOB : Lecturer and PhD Student

PHONE : 05072325511



### INFORMED VOLUNTARY CONSENT FORM

Document Code: ÜNV-GOAEK-FRM-002

Release Date: 17.09.2019

Revision No: 03

Revision Date: 01.06.2022


# **CONSENT TO PARTICIPATE IN THE STUDY**

I discussed the above information in detail with the relevant researcher and he answered all my questions. I have read and understood this informed consent document. I agree to participate in this research and sign this certificate of approval of my own free will. This approval does not invalidate any applicable laws and regulations. The researcher handed over a copy of this document to me for safekeeping.

| Volunteer Name Surname | Date and |
|-------------------------|-----------|
| | Signature |
| Phone | |
| Guardiyan (if any) Name | Date and |
| Surname | Signature |
| Phone | |
| Interview Witness Name | Date and |
| Surname | Signature |
| Phone | |
| Researcher Name Surname | Date and |
| | Signature |
| Phone | |